CLINICAL TRIAL: NCT04510272
Title: Aloud Real-time Reading of ICU Diaries for Prevention of Negative Post-ICU Psychological Outcomes: A Feasibility Study
Brief Title: Aloud Real-time Reading of ICU Diaries for Prevention of Negative Post-ICU Psychological Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Lioudmila Karnatovskaia, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-002275
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Anxiety; Depression; PTSD
Keywords: Critical illness; PTSD; Depression; anxiety; PICS
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High risk critically ill patients (Experimental): Critically ill patients requiring vasopressor support or mechanical ventilation will receive aloud real time ICU diary reading intervention
  Interventions: Other: Aloud Real-time Reading of ICU Diaries

INTERVENTIONS:
Other: Aloud Real-time Reading of ICU Diaries — Standard ICU diaries will be read aloud in real time daily to patients by ICU nurses/therapists/family members

SUMMARY:
This study will evaluate whether a systematically delivered, patient-oriented real time communication via aloud real time readings of ICU diary entries during patient's ICU stay is feasible

DETAILED DESCRIPTION:
Survivors of sepsis and acute respiratory failure suffer from long-term impairment in the domains of physical, cognitive, and psychological functioning collectively known as post intensive care syndrome (PICS) associated with increased re-hospitalization rates, higher health care costs and impaired quality of life. Pioneering work in the field of early physical rehabilitation of intensive care unit (ICU) patients and in identification of strategies for delirium reduction demonstrated improvement in physical and cognitive outcomes. Prevention of psychological complications, however, has not been adequately addressed. Anxiety, depression and post-traumatic stress disorder (PTSD) affect over a third of all critical illness survivors post discharge, which is more than double of what has been reported in combat veterans. Despite the staggering rates of mental health morbidity, research on targeting preventive measures to be employed in the ICU before development of psychological symptoms has earned sparse attention. Memories of frightening and delusional experiences appear to be the strongest potentially modifiable risk factor, with higher rates of PTSD reported in those who had delusional memories without recall of factual events. Indeed, psychiatric symptoms such as anxiety, depression, and PTSD can be conceptualized as disorders of memory content, whereby the neural representation of the emotional component of the memory of a traumatic experience persists beyond any adaptive purpose. This causes dysregulation in the fear memory system, resulting in pathology associated with impaired cognitive, affective, and volitional functions. Research on the formation of fear memories demonstrates that one can interfere with the initial process of fear conditioning during the temporal windows when memory consolidation and reconsolidation occur.

Therefore, a potential approach to treatment may be to introduce mitigating/factual information during the time period when the consolidation of the initial memory occurs and also following its initial recall, because at this time memories are labile and susceptible to alteration; however, the longer a memory has been stored in the brain, the more difficult it is to destabilize and alter it, explaining the lack of effectiveness of outpatient interventions. For the critically ill this would mean introducing some form of communication as soon as feasible following admission and providing communication in parallel with medical care in the ICU. Even though semantic processing continues in an altered states of consciousness, very little verbal communication systematically takes place with sedated and/or cognitively altered patients during the time window when the negative memories are being formed. How can such communication be introduced?

A lot of patients receive ICU diaries following hospital discharge. The original design that has remained unchanged on over 30 years has care team and family members write entries of the patient's daily events, written in a non-medical language. Despite decades of research, ICU diaries failed to demonstrate consistent benefit for mental health outcomes. What if the reason is simply due to the timing of the information provided? What is reading the entries in real time, as the events unfold, can provide that protective factual information to mitigate formation of traumatic memories?

The investigators hypothesize that reading ICU diary entries aloud in real time (in addition to providing them to patients following hospital discharge as has been the standard previously) is feasible and may translate into improved mental health outcomes including symptoms of anxiety, depression, and PTSD as well as more delirium free days. Doing so systematically may mitigate formation of false negative memories, provide reorientation and factual information, and thus help patients understand what is happening to them in real time.

This will be accomplished via the following aim:

Specific Aim #1: To conduct a feasibility trial of reading ICU diaries aloud daily and to refine the intervention based on stakeholder feedback Objective 1: ICU diaries will be read aloud in real time daily to 30 enrolled patients by ICU nurses/therapists. The approach will subsequently be refined based on semi-structured interviews of all involved stakeholders (patients, families, nurses, therapists). Patients will also complete anxiety, depression, acute stress/PTSD and cognitive function evaluation as measured by validated instruments.

ELIGIBILITY:
Inclusion Criteria:

* High risk critically ill patients: adults (age ≥ 18) in acute respiratory failure and/or requiring vasopressors admitted to the ICU and expected to stay >48 hours. adults (age ≥ 18) in acute respiratory failure and/or requiring vasopressors admitted to the ICU and expected to stay >48 hours
* Enrolled patient's family members.
* Critical care nurses.
* Physical/Occupational therapists writing ICU diary entries.

Exclusion Criteria:

* History of dementia, mental retardation, suicide attempt, psychotic disorders such as schizophrenia, acute alcohol/substance intoxication or withdrawal, severe metabolic encephalopathy; patients on comfort care; patients not expected to survive the hospital stay or non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Number of days patients successfully receive the intervention | Length of ICU admission
  Feasibility of the intervention as defined by ICU diary entries being read aloud on >80% of days they were entered

CONTACTS AND LOCATIONS:
Overall Officials: Lioudmila V Karnatovskaia, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson KR, Temeyer JP, Schulte PJ, Nydahl P, Philbrick KL, Karnatovskaia LV. Aloud real- time reading of intensive care unit diaries: A feasibility study. Intensive Crit Care Nurs. 2023 Jun;76:103400. doi: 10.1016/j.iccn.2023.103400. Epub 2023 Jan 25. PMID 36706496
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials